CLINICAL TRIAL: NCT02288429
Title: Evaluation of Steady-state Pharmacokinetic and Pharmacodynamic Properties of Intravenous Colistimethate Sodium in Cystic Fibrosis and Critically Ill Patients
Brief Title: Evaluation of Pharmacokinetic and Pharmacodynamic Properties of Intravenous Colistimethate Sodium
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2597
Record Dates: First submitted 2014-09-15; First posted 2014-11-11 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Colistin
Keywords: pharmacokinetics; cystic fibrosis; critical illness
MeSH Terms: conditions — Cystic Fibrosis; Critical Illness | interventions — colistinmethanesulfonic acid; Colistin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Colistin: * Patients ≥ 18 years old receiving intravenous colistimethate sodium for the treatment of infection
  * Have cystic fibrosis and/or are critically ill (admitted to a critical care unit)
  Interventions: Drug: colistimethate sodium

INTERVENTIONS:
Drug: colistimethate sodium
  Other Names: colistin; CMS

SUMMARY:
Colistin is a polymixin antibiotic used in the treatment of multidrug-resistant gram-negative infections. Given the limited use of colistin and previous challenges with laboratory assays to determine plasma concentrations, there is a lack of knowledge of the pharmacokinetic profile of colistin. The purpose of the investigators observational prospective pharmacokinetic cohort study is to examine the steady-state pharmacokinetic and pharmacodynamic properties of intravenous colistimethate sodium in cystic fibrosis and critically ill patients.

DETAILED DESCRIPTION:
Colistin, also known as polymixin E, is a peptide antibiotic that demonstrates concentration-dependent bactericidal killing against gram-negative pathogens including Pseudomonas and Acinetobacter. Originally discovered in the 1950s, its use has been limited due to the concern for its systemic toxicities including nephrotoxicity and neurotoxicity. However, a revival of colistin use has been seen in recent years due to the increased emergence of multidrug-resistant (MDR) gram-negative pathogens and a lack of alternative antimicrobial therapies.

Colistin is administered intravenously as colistimethate sodium (CMS), an inactive prodrug that lacks antibacterial activity, and is hydrolyzed into its active form in plasma as colistin A and colistin B. Prior pharmacokinetic studies have demonstrated a wide range of pharmacokinetic/pharmacodynamics (PK/PD) findings for colistin. Variability in results have been attributed to an unreliable differentiation between colistin and CMS plasma concentrations with the use of microbiological assays, in addition to procedures that resulted in substantial in vitro hydrolysis of CMS to colistin during sample preparation. Refined laboratory methods such as high-performance liquid chromatography (HPLC) have circumvented such issues and provided opportunities for further pharmacokinetic profiling.

Given the scarcity of its use and challenges with quantitative assays, the pharmacokinetic and pharmacodynamic profile of colistin has been poorly characterized particularly amongst cystic fibrosis and critically ill patients. Determination of such parameters in these patient populations is vital to optimize the maximum concentration to minimum inhibitory concentration (Cmax:MIC) ratio for maximal efficacy, minimize adverse effects and to reduce the development of bacterial resistance. Previous studies examining the steady-state pharmacokinetics of colistin in cystic fibrosis and critically ill patients have concluded that based on the in vitro pharmacodynamics against Pseudomonas aeruginosa, current dose recommendations may be inadequate to achieve desirable Cmax:MIC ratios and dose escalations may be warranted.

The investigators study aims to determine steady-state colistin A and colistin B concentrations in cystic fibrosis and critically ill patients, evaluate pharmacodynamic parameters and relationship to microbiologic success, and monitor for the incidence of nephrotoxicity. The findings of this pilot study will be used to develop dosing recommendations for future pharmacokinetic studies of colistimethate sodium in cystic fibrosis and critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old receiving intravenous colistimethate sodium for the treatment of infection
* Have cystic fibrosis and/or are critically ill (admitted to a critical care unit)

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at the University of Colorado Hospital
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC0-24) | 0, 30, 60, 120, 240, and 360 minutes after the IV infusion
  Steady-state plasma concentrations will be obtained after at least 2 days of therapy. Blood draws (5 ml) will be taken just before the start of the colistimethate sodium infusion and at 30, 60, 120, 240, and 360 minutes after the IV infusion.

SECONDARY OUTCOMES:
Number of patients experiencing nephrotoxicity | Baseline, during colistin therapy course (expected to be approximately 14 days), and until hospital discharge (participants will be followed for the duration of hospital stay, expected to be 2-4 weeks)
  Nephrotoxicity defined as either 1) a rise in serum creatinine (SCr) > or = 0.5 mg/dl; 2) 50% increase in SCr or 3) 25% decrease in estimated creatinine clearance

OTHER OUTCOMES:
Number of patients experiencing neurotoxicity | Baseline, during colistin therapy course (expected to be approximately 14 days), and until hospital discharge (participants will be followed for the duration of hospital stay, expected to be 2-4 weeks)
  Neurotoxicity (headache, dizziness, weakness, facial and peripheral paresthesia, vertigo, visual disturbances, confusion, ataxia, and neuromuscular blockade, or other central nervous system related symptoms) as determined by patient report

CONTACTS AND LOCATIONS:
Overall Officials: Ty Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landman D, Georgescu C, Martin DA, Quale J. Polymyxins revisited. Clin Microbiol Rev. 2008 Jul;21(3):449-65. doi: 10.1128/CMR.00006-08. PMID 18625681
- [Background] Karnik ND, Sridharan K, Jadhav SP, Kadam PP, Naidu RK, Namjoshi RD, Gupta V, Gore MS, Surase PV, Mehta PR, Gogtay JA, Thatte UM, Gogtay NJ. Pharmacokinetics of colistin in critically ill patients with multidrug-resistant Gram-negative bacilli infection. Eur J Clin Pharmacol. 2013 Jul;69(7):1429-36. doi: 10.1007/s00228-013-1493-9. Epub 2013 Mar 19. PMID 23508665
- [Background] Plachouras D, Karvanen M, Friberg LE, Papadomichelakis E, Antoniadou A, Tsangaris I, Karaiskos I, Poulakou G, Kontopidou F, Armaganidis A, Cars O, Giamarellou H. Population pharmacokinetic analysis of colistin methanesulfonate and colistin after intravenous administration in critically ill patients with infections caused by gram-negative bacteria. Antimicrob Agents Chemother. 2009 Aug;53(8):3430-6. doi: 10.1128/AAC.01361-08. Epub 2009 May 11. PMID 19433570
- [Background] Li J, Coulthard K, Milne R, Nation RL, Conway S, Peckham D, Etherington C, Turnidge J. Steady-state pharmacokinetics of intravenous colistin methanesulphonate in patients with cystic fibrosis. J Antimicrob Chemother. 2003 Dec;52(6):987-92. doi: 10.1093/jac/dkg468. Epub 2003 Oct 29. PMID 14585859
- [Background] Ratjen F, Rietschel E, Kasel D, Schwiertz R, Starke K, Beier H, van Koningsbruggen S, Grasemann H. Pharmacokinetics of inhaled colistin in patients with cystic fibrosis. J Antimicrob Chemother. 2006 Feb;57(2):306-11. doi: 10.1093/jac/dki461. Epub 2006 Jan 5. PMID 16396919
- [Background] Markou N, Markantonis SL, Dimitrakis E, Panidis D, Boutzouka E, Karatzas S, Rafailidis P, Apostolakos H, Baltopoulos G. Colistin serum concentrations after intravenous administration in critically ill patients with serious multidrug-resistant, gram-negative bacilli infections: a prospective, open-label, uncontrolled study. Clin Ther. 2008 Jan;30(1):143-51. doi: 10.1016/j.clinthera.2008.01.015. PMID 18343250
- [Background] Imberti R, Cusato M, Villani P, Carnevale L, Iotti GA, Langer M, Regazzi M. Steady-state pharmacokinetics and BAL concentration of colistin in critically Ill patients after IV colistin methanesulfonate administration. Chest. 2010 Dec;138(6):1333-9. doi: 10.1378/chest.10-0463. Epub 2010 Jun 17. PMID 20558557